CLINICAL TRIAL: NCT03148249
Title: A Randomized Control Trial of Patients With a Charles Bonnet Syndrome
Brief Title: A Trial of Patients With a Charles Bonnet Syndrome
Acronym: CBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Univ. Prof. Dr., MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIROS
Record Dates: First submitted 2017-02-09; First posted 2017-05-10 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Prevalence, Psychiatrist Intervention
Keywords: Randomized control trial; Charles Bonnet syndrome; visual hallucinations; age related macular degeneration; patient education
MeSH Terms: conditions — Charles Bonnet Syndrome; Hallucinations; Macular Degeneration | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interview with an ophthalmologist (Experimental): Patients get an interview with an ophthalmologist
  Interventions: Other: interview
- interview/treatment by a psychiatrist (Experimental): patients get an interview and a possible treatment by a psychiatrist
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — control group: interview, study group: explanation and exploration

SUMMARY:
Charles Bonnet Syndrome (CBS) is defined by the occurence of visual hallucinations (VH) in the absence of any mental disorder. Elderly patients with reduced visual acuity due to ophthalmic diseases are most affected. Conditions are often associated with the syndrome of age-related macular degeneration, cataract or glaucoma. Existing data on the syndrome's prevalence in Europe reveal diverse results. Aim of this study was to assess the prevalence of CBS in patients with low visual acuity and to evaluate, if an additional therapeutic interview with and treatment by a psychiatrist is beneficial.

DETAILED DESCRIPTION:
Patients with a visual acuity of 0.5 LogMAR or less in the better eye were screened for CBS. Instruments used were an interview asking for details of the hallucinations, a mental test and a scale concerning quality of life. Patients with CBS were randomized by minimization in two groups: in group 1, a patient-doctor interview by an ophthalmologist was performed and in group 2 an interview and if needed, a therapy by a psychiatrist. At the 3-months follow up, the psychological strain of patients was recorded again.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* visual acuity of 0.5 LogMAR or less at both eyes
* 55 years or older

Patients with CBS:

* have no mental pathologies such as dementia, psychosis or any other neurological diseases
* have a normal cognitive state
* are not able to control the VH
* know that the VH are not real
* are usually older
* have significantly reduced visual acuity due to an bilateral eye pathology

VH associated with CBS:

* disappear when the eyes are closed
* are repetitive
* are complex (eg. objects, geometrical patterns, faces, shapes, figures, scenes, animals or plants)

Exclusion Criteria:

* dopamine agonist medication
* temporal lobe epilepsy
* moderate to severe Alzheimer's dementia
* present chronic alcohol-/drug abuse
* bad cognitive state

There are no:

* auditory or olfactory hallucinations
* other abnormalities like delusions

Ages: 55 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Quality of life score between the two groups | 3 months
  Quality of life score between the study and control group

IPD SHARING:
Plan to Share IPD: No